CLINICAL TRIAL: NCT04804891
Title: Using T-Cell Alloreactivity and Chimerism to Guide Immunosuppression Minimization in Intestinal Transplantation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Ossium Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAS8908
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Intestinal Transplantation
Keywords: CD34+ stem cells; Chimerism; Bone marrow stells
MeSH Terms: interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cell Therapy (Experimental): Patients will receive an infusion containing 1x106/kg CD34+ cells. No more than 104 CD34+ T cells per kg recipient weight will be included in the infusion. Cadaveric donor CD34 cell infusion will occur at any time between post-operative day 11 to day 13 following transplantation.
  Interventions: Biological: Cell Therapy
- Control (No Intervention): Patients who do not consent to receive donor CD34 cell infusion or whose donor family declines consent for research use of donor bone marrow will receive their usual standard of care.

INTERVENTIONS:
Biological: Cell Therapy — Infusion of containing 1x106/kg CD34+ cells from donor bone marrow selected using the CliniMACS® CD34 Reagent System.
  Arms: Cell Therapy

SUMMARY:
The purpose of this study is to investigate the safety and feasibility of giving intestinal transplant patients CD34+ stem cells (the cells that make all the types of blood cells) obtained from their organ donor's bone marrow. The goal of this is to develop a post-transplant treatment strategy that controls rejection while reducing the high risk of infection and malignant disease associated with the high levels of immunosuppression medication(s) that intestinal and multi-organ transplant patients must take. Infusion of bone marrow cells from the same donor of the transplanted organ(s) could promote a state called "mixed chimerism" in which both donor cells and recipient cells coexist in the body with the ultimate goal of minimizing the amount of immunosuppression medication(s) needed.

DETAILED DESCRIPTION:
Abdominal trauma, congenital abnormalities and ischemic injury cause intestinal damage that prevents the digestion and absorption of fluids and nutrients essential for life. Intestinal transplantation is life-saving for patients with complications related to the administration of intravenous nutrients. Approximately 100-160 intestinal transplants (ITx) are performed in the US annually. However, patient survival rates are far from optimal, due to high rejection rates resulting from an immune attack of the recipient against the donor, termed host-vs-graft (HVG) reactivity The high levels of global immunosuppression used to prevent rejection come with a high risk of infections and malignant disease (i.e. lymphoma). Thus, there is an urgent need for a well-tolerated treatment strategy that controls rejection while reducing these risks. Immune tolerance, in which the immune system regards the donor as "self" so that long-term graft acceptance is achieved without life-long immunosuppression, would accomplish this goal . Infusion of bone marrow cells from the same donor of the solid organs could promote a state called "mixed chimerism" in which both donor cells and recipient cells coexist in the body. Mixed chimerism has been shown to induce tolerance to the transplanted organ in animal models and in patients receiving kidney transplants.

The investigators propose studies to promote tolerance induction in intestinal transplant recipients by administering donor bone marrow stem cells to promote lasting mixed chimerism. The investigators' proposal builds on their demonstration that mixed chimerism commonly occurs in intestinal transplant (ITx) recipients without bone marrow transplant, and that its presence correlates with reduced rejection rates. However, this mixed chimerism is not permanent. The investigators have discovered that there are bone marrow stem cells in the donor intestinal grafts and that some of these survive and enter the bone marrow of the recipient. This process is facilitated by a phenomenon called a "lymphohematopoietic graft-vs-host responses (LGVHR)", in which T lymphocytes from the ITx donor attack recipient blood-forming cells to make "space" for their own establishment in the bone marrow, but do not induce GVHD. The investigators have also obtained evidence that this immune response suppresses rejection of the graft.

ELIGIBILITY:
Inclusion Criteria:

* All patients actively listed as candidates for intestinal or multi-visceral transplant at the study site; while all patients who are actively listed in United Network for Organ Sharing (UNOS) for intestinal and/or multi-visceral transplantation, including those who have previously received a multi-visceral transplant and are re-listed, are eligible for participation, the following are examples of listing criteria suitable for enrollment in this clinical trial:

  * Short Bowel Syndrome (SBS) due to:

    * Trauma (multiple resections/explorations and/or vascular abdominal trauma superior mesenteric artery (SMA) / superior mesenteric vein (SMV) injuries)
    * Gastroschisis
    * Volvulus
    * Necrotizing Enterocolitis
    * Intestinal Atresia
    * Crohn's Disease
    * Hirschprung's Disease
  * Chronic Intestinal Pseudo-Obstruction
  * Malabsorption:

    * Microvillus Inclusion Disease
    * Tufting Enteropathy
    * Complete portomesenteric thrombosis with cirrhosis
  * Slow-growing, low-malignancy potential tumors infiltrating mesenteric root:

    * Gardner's Syndrome
    * Familial Adenomatous Polyposis
    * Desmoid Tumor with Intra-Abdominal Infiltration
    * Endocrine Tumors
  * Re-transplant candidates who lost the first graft to rejection or patients who have higher risk of toxicity from chronic long term immunosuppression (i.e., patients with chronic kidney disease)
* Patient commits to planned follow up at a study site for the 48-month duration of study procedures
* Age ≥18 years old and ≤65 years old
* Subjects or capable of signing the informed consent document themselves

Exclusion Criteria:

* Active systemic infection with hemodynamic instability and/or sepsis
* Patients with known immunodeficiency syndrome
* Carcinoma with metastasis (except neuro-endocrine tumors, even in the presence of metastasis these patients may undergo multivisceral/cluster transplantation)
* Severe cardiovascular and/or respiratory instability, as defined by requirement of pressors or ventilator
* Severe cerebral edema, with radiologic findings of effaced sulci and/or herniation
* Poorly controlled hypertension (systolic blood pressure > 170 on at least 2 occasions), diabetes mellitus (HbA1c > 8), or uncontrollable seizure disorders
* Age > 65 years
* Documented history of non-compliance with medical therapy and follow-up
* Substance addiction in the last six months
* Psychosocial Instability: absence of a consistent reliable social support system
* Significant or active psychiatric disorder associated with the inability to cooperate or comply with medical therapy
* In the judgement of the clinical team, severely limited functional status with poor rehabilitation potential
* Multi-organ failure and preceding CD34+ infusion
* Pre formed panel reactive antibodies (PRA) mean fluorescein intensity (MFI) > 5000 by Luminex
* Patients who are pregnant or breast-feeding or intend to get pregnant during the study period
* Patients who have developed moderate or severe rejection before post-transplant day 11
* Vulnerable populations, such as incarcerated or institutionalized individuals
* Subjects with clinical features suggestive of GVHD
* Subjects who are hemodynamically unstable (i.e., requiring vasopressor support)
* Female subjects of childbearing age and male patients who are not using and/or unwilling to use an effective method of birth control for the duration of the trial activities
* History of previous hematopoietic progenitor cell (HPC) infusion or transplant of any kind. Note: Human leukocyte antigen (HLA) mismatch will not be one of the exclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Total number of participants with moderate to severe GVHD | Up to 4 years after transplantation
  Total number of participants with moderate to severe (at least Grade II) graft-versus-host disease (GVHD) will be monitored.

SECONDARY OUTCOMES:
Graft survival rate | Up to 1 month after transplantation
  Percentage of individuals with graft survival.
Retention rate | Up to 1 month after transplantation
  Percentage of individuals with retention from any cause.
Graft survival rate | Up to 1 year after transplantation
  Percentage of individuals with graft survival.
Retention rate | Up to 1 year after transplantation
  Percentage of individuals with retention from any cause.
Graft survival rate | Up to 3 years after transplantation
  Percentage of individuals with graft survival.
Retention rate | Up to 3 years after transplantation
  Percentage of individuals with retention from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Tomoaki Kato, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/NYP, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided